CLINICAL TRIAL: NCT04977401
Title: EndoscoPic Submucosal dIssection Using geL Versus glycerOl for Submucosal iNjection: a Randomized Controlled Multicentric Trial (EPSILON)
Brief Title: EndoscoPic Submucosal dIssection Using geL Versus glycerOl for Submucosal iNjection
Acronym: EPSILON
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Urgent Medical Device Product (ORISE Gel Submucosal Liftiong Agent) Removal by sponsor
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Lemmers Arnaud, MD, PhD, Professor, Head of Clinic, Endoscopy Unit, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPSILON
Record Dates: First submitted 2021-07-08; First posted 2021-07-26 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Early Gastric Cancer; Rectal Polyp
Keywords: ESD (endoscopic submucosal dissection); Rectum polyp; early gastric cancer; endoscopic resection; submucosal injection solution
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Intervention Model Description: A multicentric, randomized, open label prospective study:
  * All subjects with indications of gastric and rectal ESD undergo screening and baseline visit
  * Informed consent is obtained when scheduling the ESD procedure
  * Randomization is made at the time of the ESD procedure after confirmation of the indication
  * ESD is performed using a 25 G needle, a dual-knife-J with glycerol (standard solution) or ORISETM gel in order to remove the lesion en-bloc. Additional saline injection through the electrosurgical knife will be left at the discretion of the endoscopist
  * A follow-up visit is scheduled at 2-4 weeks
Who Masked: Participant
Masking Description: A computer-based block randomization scheme will be created using block randomization and stratifying by center and by organ type (stomach/rectum). Data will be collected through a printed CRFs and then anonymized and entered into a central web based secured platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Glycerol (Sham Comparator): Submucosal injection using glycerol during an ESD procedure in a specific population with superficial gastric and rectal (pre)neoplastic lesions.
  Interventions: Procedure: Endoscopic submucosal dissection; Device: use of glycerol as lifting agent for endoscopic submucosal dissection
- Group Gel ORISE (Active Comparator): Submucosal injection using ORISETM gel during an ESD procedure in a specific population with superficial gastric and rectal (pre)neoplastic lesions.
  Interventions: Procedure: Endoscopic submucosal dissection; Device: use of Orise Gel as lifting agent for endoscopic submucosal dissection

INTERVENTIONS:
Procedure: Endoscopic submucosal dissection — Dissecting superficial gastric or rectal lesion/polyp after injection of the submucosa for lifting, using a electrosurgical knife through the endoscope
Device: use of Orise Gel as lifting agent for endoscopic submucosal dissection — Injection of some colloidal solution (ORISE gel) in the submucosal layer in order to obtain long lifting effect and thus allowing the endoscopist to dissect under the lesion.
  Arms: Group Gel ORISE
Device: use of glycerol as lifting agent for endoscopic submucosal dissection — Injection of some colloidal solution (glycerol) in the submucosal layer in order to obtain long lifting effect and thus allowing the endoscopist to dissect under the lesion.
  Arms: Group Glycerol

SUMMARY:
The EPSILON study aims to comparatively evaluate the submucosal injection using ORISETM gel and glycerol during an ESD procedure in a specific population with superficial gastric and rectal (pre)neoplastic lesions.

DETAILED DESCRIPTION:
Traditionally, ESD requires the injection of some colloidal solution (glycerol, geloplasma, hydroxyethylstrach, etc.) in the submucosal layer in order to obtain long lifting effect and thus allowing the endoscopist to dissect under the lesion. Alternatives to colloid-solution assisted ESD have also been developped: pocket creation method and saline-immersion ESD.

Recently, other colloidal solutions have arrived on the market, such as gel (ORISETM gel) in order to improve the lifting during ESD.Our preliminary experience using ORISETM gel as a lifting solution for ESD was unexpectedly favourable with few per-procedural bleeding, quick time and facility.

As the spread of ESD is closely associated to its easiness, procedure duration (itself associated to number of procedural bleedings and instruments change through the operating channel) and safety, we sought to study comparatively two submucosal solutions when conducting ESD in a specific population presenting gastric or rectal superficial lesions.

ELIGIBILITY:
Inclusion Criteria:

* o Patients must have given written informed consent
* o Subjects with documented gastric or rectal lesions with indication of endoscopic removal by ESD, namely:

  * Gastric focal lesion with suspicion of early gastric cancer (low or high grade dysplasia with features of early gastric cancer; adenocarcinoma with morphology of superficial lesion and work-up of superficial lesion)
  * Rectal polyps (adenoma or superficial carcinoma) from 0 to 15 cm from the anal margin; with features being recognized indications of ESD: more than 20mm granular LST, more than 20mm non granular LST, more than 20mm villous or bulging polyps, Paris 0-IIa+IIc lesions, lesions with suspicious pattern (Kudo Vi / JNET 2B), lesions with anal canal involvement.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria cannot be enrolled in the study:

  * Gastric and rectal neuroendocrine tumour (NET) with indication of ESD will be excluded
  * Gastric and rectal lesions with indication of ESD but strong fibrosis due to previous partial resection will be excluded
  * Subject is currently enrolled in another confounding research
  * Subjects with any other location of ESD (esophagus, duodenum and colon) will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Increase the dissection speed of the ESD procedure | At day 0 during ESD
  Increase the dissection speed of the ESD procedure (defined as the dissected surface (mm2)/ESD duration (min). The dissected surface is defined as maximal diameter of specimen (mm) x perpendicular minimal diameter of specimen (mm) measured on ex-vivo pinned stretched specimen onto a cork. ESD duration is defined as the time from first submucosal injection to final cut time.

SECONDARY OUTCOMES:
Total procedure duration | At day 0 during ESD
  Total procedure duration (from scope insertion to scope retrieval) (min)

OTHER OUTCOMES:
Number of per-procedural bleeding | At day 0 during ESD
  Number of per-procedural bleeding (+ severity scale: oozing / severe non pulsating/ severe pulsating)
Total hemostatic time | At day 0 during ESD
  Total hemostatic time (addition of each hemostasis time for each per-procedural bleeding)
Need for haemostatic forceps | At day 0 during ESD
  Need for haemostatic forceps during ESD
Difficulty of the dissection | At day 0 during ESD
  Difficulty of the dissection (scale) (very easy / easy / moderately difficult / difficult / very difficult)
Amount of submucosal solution | At day 0 during ESD
  Amount of submucosal solution (glycerol or gel) used for ESD in ml
Combined use of saline | At day 0 during ESD
  Combined use of saline through the knife during ESD (number and ml)
Number of needle injection dots | At day 0 during ESD
  Number of needle injection dots during ESD (initially / during ESD)
Need to adjust electrosurgical settings | At day 0 during ESD
  Need to adjust electrosurgical settings during ESD
Clear visualisation of the plane of dissection during ESD (scale). | At day 0 during ESD
  Clear visualisation of the plane of dissection during ESD (scale). The scale will be defined according the endoscopists evaluation of the delineation between the submucosa ad the underlying muscular layer:
  * Very-good visualization: clear delineation between the two layers with clear visualization of the blood vessels.
  * Good visualization: mostly clear delineation between the two layers, but with blurred regions
  * Bad visualization: delineation between the two layers is unclear (i.e.:
  fibrosis)
Rate of en-bloc dissection | At day 0 during ESD
  Rate of en-bloc dissection (defined as endoscopic resection of the targeted area in one bloc)
Rate of complete endoscopic resection | At day 0 during ESD
  Rate of complete endoscopic resection (defined as endoscopic evaluation of complete removal of the targeted area in the treated organ)
Quality assessment of the pathological specimen | At day 0 during ESD
  Quality assessment of the pathological specimen (absolute measure of the depth of resected submucosa on the specimen, rate of clear (horizontal and vertical) margins)
Adverse events | From ICF signature up to 2-3 weeks follow-up
  Adverse events:
  * Per-procedural (incidence of all adverse technical events during the procedure)
  * Early (clinical and laboratory at 24 h post procedure according to CTCAE v 5.0)
  * Late (clinical at 2-3 weeks follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Lemmers, MD,PhD, Principal Investigator — Erasme Hospital, Université Libre de Bruxelles. (ULB), Brussels, Belgium
Locations (3):
- Erasme Hospital, Université Libre de Bruxelles. (ULB), Brussels, Belgium
- Evangelisches Krankenhaus, Düsseldorf, Germany
- Keio University Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao Y, Liao C, Tan A, Gao Y, Mo Z, Gao F. Meta-analysis of endoscopic submucosal dissection versus endoscopic mucosal resection for tumors of the gastrointestinal tract. Endoscopy. 2009 Sep;41(9):751-7. doi: 10.1055/s-0029-1215053. Epub 2009 Aug 19. PMID 19693750
- [Result] Fujishiro M. Perspective on the practical indications of endoscopic submucosal dissection of gastrointestinal neoplasms. World J Gastroenterol. 2008 Jul 21;14(27):4289-95. doi: 10.3748/wjg.14.4289. PMID 18666315
- [Result] Kodashima S, Fujishiro M, Yahagi N, Kakushima N, Omata M. Endoscopic submucosal dissection using flexknife. J Clin Gastroenterol. 2006 May-Jun;40(5):378-84. doi: 10.1097/00004836-200605000-00004. PMID 16721217
- [Result] Park YM, Cho E, Kang HY, Kim JM. The effectiveness and safety of endoscopic submucosal dissection compared with endoscopic mucosal resection for early gastric cancer: a systematic review and metaanalysis. Surg Endosc. 2011 Aug;25(8):2666-77. doi: 10.1007/s00464-011-1627-z. Epub 2011 Mar 18. PMID 21424201
- [Result] Lian J, Chen S, Zhang Y, Qiu F. A meta-analysis of endoscopic submucosal dissection and EMR for early gastric cancer. Gastrointest Endosc. 2012 Oct;76(4):763-70. doi: 10.1016/j.gie.2012.06.014. Epub 2012 Aug 9. PMID 22884100
- [Result] Pimentel-Nunes P, Dinis-Ribeiro M, Ponchon T, Repici A, Vieth M, De Ceglie A, Amato A, Berr F, Bhandari P, Bialek A, Conio M, Haringsma J, Langner C, Meisner S, Messmann H, Morino M, Neuhaus H, Piessevaux H, Rugge M, Saunders BP, Robaszkiewicz M, Seewald S, Kashin S, Dumonceau JM, Hassan C, Deprez PH. Endoscopic submucosal dissection: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2015 Sep;47(9):829-54. doi: 10.1055/s-0034-1392882. Epub 2015 Aug 28. PMID 26317585
- [Result] Fujishiro M, Yahagi N, Kashimura K, Mizushima Y, Oka M, Enomoto S, Kakushima N, Kobayashi K, Hashimoto T, Iguchi M, Shimizu Y, Ichinose M, Omata M. Comparison of various submucosal injection solutions for maintaining mucosal elevation during endoscopic mucosal resection. Endoscopy. 2004 Jul;36(7):579-83. doi: 10.1055/s-2004-814517. PMID 15243878
- [Result] Castro R, Libanio D, Pita I, Dinis-Ribeiro M. Solutions for submucosal injection: What to choose and how to do it. World J Gastroenterol. 2019 Feb 21;25(7):777-788. doi: 10.3748/wjg.v25.i7.777. PMID 30809079
- [Result] Takezawa T, Hayashi Y, Shinozaki S, Sagara Y, Okada M, Kobayashi Y, Sakamoto H, Miura Y, Sunada K, Lefor AK, Yamamoto H. The pocket-creation method facilitates colonic endoscopic submucosal dissection (with video). Gastrointest Endosc. 2019 May;89(5):1045-1053. doi: 10.1016/j.gie.2019.01.022. Epub 2019 Feb 1. PMID 30716306
- [Result] Yamamoto H, Hayashi Y, Despott EJ. The pocket-creation method for endoscopic submucosal dissection combined with saline-immersion: another potential option to overcome challenges in colorectal endoscopic submucosal dissection. Gastrointest Endosc. 2019 Aug;90(2):288-289. doi: 10.1016/j.gie.2019.04.244. No abstract available. PMID 31327340
- [Result] Endoscopic Classification Review Group. Update on the paris classification of superficial neoplastic lesions in the digestive tract. Endoscopy. 2005 Jun;37(6):570-8. doi: 10.1055/s-2005-861352. PMID 15933932
- [Result] Hewett DG, Kaltenbach T, Sano Y, Tanaka S, Saunders BP, Ponchon T, Soetikno R, Rex DK. Validation of a simple classification system for endoscopic diagnosis of small colorectal polyps using narrow-band imaging. Gastroenterology. 2012 Sep;143(3):599-607.e1. doi: 10.1053/j.gastro.2012.05.006. Epub 2012 May 15. PMID 22609383
- [Result] Sano Y, Tanaka S, Kudo SE, Saito S, Matsuda T, Wada Y, Fujii T, Ikematsu H, Uraoka T, Kobayashi N, Nakamura H, Hotta K, Horimatsu T, Sakamoto N, Fu KI, Tsuruta O, Kawano H, Kashida H, Takeuchi Y, Machida H, Kusaka T, Yoshida N, Hirata I, Terai T, Yamano HO, Kaneko K, Nakajima T, Sakamoto T, Yamaguchi Y, Tamai N, Nakano N, Hayashi N, Oka S, Iwatate M, Ishikawa H, Murakami Y, Yoshida S, Saito Y. Narrow-band imaging (NBI) magnifying endoscopic classification of colorectal tumors proposed by the Japan NBI Expert Team. Dig Endosc. 2016 Jul;28(5):526-33. doi: 10.1111/den.12644. Epub 2016 Apr 20. PMID 26927367

DOCUMENTS (2):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT04977401/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT04977401/SAP_001.pdf